CLINICAL TRIAL: NCT00478569
Title: Adherence to PTH(1-84) Treatment in Europe. A Non-interventional Cohort Study Collecting Safety Information and Examining Reasons and Predictors for Adherence to PTH(1-84) Treatment in Usual Clinical Settings
Brief Title: Adherence to PTH(1-84) Treatment (FP-002-IM)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: FP-002-IM
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-04

CONDITIONS: Clinical Use of PTH(1-84)
MeSH Terms: interventions — Parathyroid Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parathyroid Hormone (PTH) (1-84): PTH(1-84) was prescribed in accordance with the terms of the marketing authorization. Participants were observed for 24 months.
  Interventions: Drug: Parathyroid Hormone (PTH) (1-84)

INTERVENTIONS:
Drug: Parathyroid Hormone (PTH) (1-84) — Adherence to PTH(1-84) treatment in Usual Clinical Settings
  Other Names: Preotact

SUMMARY:
The primary objective is:

1) to describe adherence (and the main factors influencing adherence) to PTH(1-84) treatment when prescribed in a normal clinical setting.

The secondary objectives are:

1. to describe the demographics and clinical characteristics of the patients that in a normal clinical setting are started on a treatment regimen with PTH(1-84)
2. to describe (using available data) the long term treatment effectiveness during the 24 months following initiation of PTH(1-84) treatment in a normal clinical setting
3. to monitor safety for 24 months following initiation of PTH(1-84) treatment in a patient in a normal clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* According to the current Summary of Product Characteristics (SmPC)
* PTH(1-84) treatment initiated within one month preceding enrolment
* The patient's written informed consent to direct access and data processing must be obtained.

Exclusion Criteria:

* According to the current SmPC
* The patient cannot participate in a clinical trial with PTH (all other trials allowed).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with osteoporosis and a high risk of fractures prescribed PTH(1-84) in a normal clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 1179 (Actual)
Dates: Start 2007-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (1):
- Nycomed, Roskilde, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 120 investigative sites in Austria, Denmark, Germany, Greece, Ireland, the Netherlands, Spain, and the United Kingdom from 1 April 2007 to 6 March 2013.
Pre-assignment Details: Participants with a diagnosis of osteoporosis and prescribed parathyroid hormone (PTH)(1-84) in a normal clinical setting were enrolled in this non-interventional study for 24 months observation. 1179 participants were enrolled however for 9 patients the data was missing.
Period: Overall Study
Arm/Group | Parathyroid Hormone (PTH) (1-84)
Started | 1170
Completed | 761
Not Completed | 409

BASELINE CHARACTERISTICS:
Arm/Group | Parathyroid Hormone (PTH) (1-84)
Number analyzed (Participants) | 1170
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (9.05)
Sex/Gender, Customized [Number; unit: participants] — Although the indication in the Summary of Product characteristics is only females, some males were initially enrolled in countries where the PTH treatment is reimbursed.
  participants
    Male | 19
    Female | 1149
    Missing | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1165
  Asian | 1
  African | 1
  Other | 1
  Missing | 2
Region of Enrollment [Number; unit: participants]
  Austria | 158
  Denmark | 79
  Germany | 246
  Greece | 300
  Ireland | 29
  Netherlands | 65
  Spain | 272
  United Kingdom | 21
Height [Mean (Standard Deviation); unit: cm] | 156.3 (7.98)
Weight [Mean (Standard Deviation); unit: kg] | 63.4 (12.25)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (4.59)
Age at Onset of Menopause [Mean (Standard Deviation); unit: years] — Total number of menopausal participants at baseline was 1148.
  years | 47.9 (5.49)
Age at Onset of Menopause by Category [Number; unit: participants] — Total number of menopausal participants at baseline was 1148, respectively.
  participants
    ≤ 45 years | 283
    > 45 years | 749
    Missing | 116
Type of Menopause [Number; unit: participants] — Total number of menopausal participants at baseline was 1148.
  participants
    Surgical | 137
    Natural | 966
    Other | 25
    Missing | 20
Calcium and/or Vitamin D Supplement [Number; unit: participants]
  Yes | 1046
  No | 122
  Missing | 2
Time Since Starting PTH(1-84) [Mean (Standard Deviation); unit: days] | 8.1 (15.52)
PTH (1-84) Dosing Frequency [Number; unit: participants]
  Once Daily | 1162
  Every Other Day | 6
  Missing | 2
Family History of Osteoporosis [Number; unit: participants]
  Yes | 223
  No | 896
  Unknown | 1
  Missing | 50
Alcohol Consumption [Number; unit: participants]
  Never | 709
  Occasionally | 385
  Daily | 50
  Missing | 26
Current Smoker [Number; unit: participants]
  Yes | 111
  No | 1057
  Missing | 2
Past Smoker [Number; unit: participants]
  Yes | 159
  No | 1009
  Missing | 2
Glucocorticosteroid Use [Number; unit: participants]
  Yes | 129
  No | 1038
  Missing | 3
Total Hip Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2] — Measured by dual energy X-ray absorptiometry (DXA). The total number of participants for whom baseline hip BMD data was available was 654.
  g/cm^2 | 0.680 (0.1239)
Total Hip T-score [Mean (Standard Deviation); unit: units on a scale] — T-score is the bone mineral density (BMD) at the site when compared to the young normal reference mean; a healthy thirty-year-old.
  Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5 Osteoporosis is defined as -2.5 or lower.
  The total number of participants for whom Baseline hip T-score data was available was 812.
  units on a scale | -2.46 (0.965)
Spine Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2] — The total number of participants for whom baseline spine bone mineral density data was available was 738.
  g/cm^2 | 0.763 (0.1480)
Spine T-score [Mean (Standard Deviation); unit: units on a scale] — The total number of participants for whom Baseline spine T-score data was available was 954.
  units on a scale | -3.10 (1.130)
Number of Participants With at Least One Fracture [Number; unit: participants] | 904
Was Patient/relative/helper instructed in PTH(1-84) (self) injection technique? [Number; unit: participants]
  Yes | 1167
  No | 1
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued Before 6 Months of Treatment
Description: A participant was defined as "permanently discontinued" if treatment with PTH(1-84) was not ongoing at the 6-month time point and at any future time points afterwards.
Time Frame: 6 months
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | Parathyroid Hormone (PTH) (1-84)
Number analyzed (Participants) | 1170
participants | 181

2. Secondary Outcome: Number of Participants Who Discontinued Before 3, 12, 18, and 24 Months of Treatment
Description: A participant was defined as "permanently discontinued" if treatment with PTH(1-84) was not ongoing at the 6-month time point and at any future time points afterwards. A participant was defined as "temporarily discontinued" if treatment with PTH(1-84) was not ongoing at the time point but was then ongoing at a future time point. This was the case when a participant or investigator wanted to pause the treatment for a length of time (e.g. because of an adverse event or interruption). Therefore, a participant was defined as still "ongoing" during the trial if treatment with PTH(1-84) had not been permanently or temporarily discontinued at that time point. A participant was only defined as "missing" or "unknown" if they attended the relevant visit and there was no result or "unknown" was entered as the result. Results for months 3, 12, 18 and 24 are cumulative data up until that time point.
Time Frame: From enrollment to 3, 12, 18, and 24 months
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | 3 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 1170 | 1170 | 1170 | 1170
participants
  Permanently discontinued | 75 | 198 | 284 | 525
  Temporarily discontinued | 6 | 8 | 2 | 2
  Ongoing | 898 | 847 | 709 | 375
  Unknown | 0 | 0 | 0 | 0
  Missing | 191 | 117 | 175 | 268

3. Secondary Outcome: Duration of Treatment
Description: Duration of treatment was defined as the last known date that PTH(1-84) was taken minus the first date that PTH(1-84) was taken plus one. In the calculation of duration, no adjustment was made for the prescribed dose frequency or for periods of temporary discontinuation due to adverse drug reactions (ADRs) or temporary patient suspension of treatment.
Time Frame: 24 months
Population: Participants for whom data were available
Measure: Mean (Full Range); unit: months
Arm/Group | Parathyroid Hormone (PTH) (1-84)
Number analyzed (Participants) | 1156
months | 17.7 [0 to 35]

4. Secondary Outcome: Treatment Compliance by Visit
Description: A participant was defined as compliant if the participant took the treatment as prescribed by the Physician, i.e. complied with the Physician's advice and followed the treatment regimen prescribed. A participant whose dose frequency and treatment length were changed during treatment, e.g. in response to a raised serum calcium level, was regarded as fully compliant if the revised treatment regimen was adhered to.
  Data on compliance were obtained at each visit and relate to the period since the previous recorded visit.
Time Frame: From enrollment to 3, 6, 12, 18, and 24 months
Measure: Number; unit: participants
Arm/Group | 3 Months | 6 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 1170 | 1170 | 1170 | 1170 | 1170
participants
  Compliant | 875 | 845 | 800 | 721 | 558
  Non-compliant | 105 | 80 | 95 | 89 | 93
  Missing | 190 | 245 | 275 | 360 | 519

ADVERSE EVENTS:
Time Frame: 24 months
Description: At each visit the investigator had to document any occurrence of adverse drug reactions and abnormal laboratory findings related to the treatment.
Arm/Group | Parathyroid Hormone (PTH) (1-84)
Serious Adverse Events (participants affected / at risk) | 10/1170
Other Adverse Events (participants affected / at risk) | 276/1170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parathyroid Hormone (PTH) (1-84) (N=1170)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Blood calcium increased (Investigations) | 1
Weight decreased (Investigations) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parathyroid Hormone (PTH) (1-84) (N=1170)
Palpitations (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 5
Motion sickness (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 5
Hyperparathyroidism (Endocrine disorders) | 1
Panophthalmitis (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 66
Reflux gastritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 1
Chills (General disorders) | 2
Discomfort (General disorders) | 1
Fatigue (General disorders) | 6
Feeling abnormal (General disorders) | 1
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site haematoma (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 9
Pain (General disorders) | 4
Pyrexia (General disorders) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Blood alkaline phosphatase increased (Investigations) | 3
Blood calcium abnormal (Investigations) | 1
Blood pressure systolic increased (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 123
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Balance disorder (Nervous system disorders) | 1
Burning sensation mucosal (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 27
Paraesthesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Hypercalciuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash papulosquamous (Skin and subcutaneous tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related publication will be multi-center or single-center publications. All proposed site publications and presentations will be submitted to (sponsor) NPS Pharmaceuticals for review in advance of publication.